CLINICAL TRIAL: NCT02272621
Title: Bleeding in Partial Upper Hemisternotomy Versus Full Sternotomy Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magnus Dalén, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMILE-bleeding
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partial upper hemisternotomy aortic valve replacement (Experimental): Partial upper hemisternotomy AVR will be performed according to current standard of care practices.
  Interventions: Procedure: Minimally invasive aortic valve replacement
- Full sternotomy aortic valve replacement (Experimental): Full sternotomy AVR through a standard median sternotomy will be performed according to current standard of care practices.
  Interventions: Procedure: Full sternotomy aortic valve replacement

INTERVENTIONS:
Procedure: Minimally invasive aortic valve replacement
  Arms: Partial upper hemisternotomy aortic valve replacement
Procedure: Full sternotomy aortic valve replacement
  Arms: Full sternotomy aortic valve replacement

SUMMARY:
This is a single-center, open-label, randomized controlled trial. Patients scheduled for aortic valve replacement (AVR) at Karolinska University Hospital in Stockholm, Sweden will be eligible. One-hundred patients will be randomly assigned to either partial upper sternotomy (50 patients) or full sternotomy AVR (50 patients). Inclusion criteria is severe aortic stenosis referred for medically indicated isolated aortic valve replacement. Exclusion criteria are inclusion in other trial, left ventricular ejection fraction less than 0.45, previous cardiac surgery, or urgent/emergent surgery.

Mechanical and bioprosthetic (stented or sutureless) aortic valves will be implanted. Clinical characteristics will be registered. Clinical postoperative outcomes including bleeding outcomes will be registered. Routine blood sampling will be performed pre- and postoperatively. All available data will be collected prospectively. Informed consent will be obtained from patients meeting the inclusion criteria before the initiation of any study-specific procedures.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Severe aortic stenosis defined as aortic valve area of less than 1 cm2 or index area of 0.6 cm2/m2 by echocardiography
* Referred for medically indicated aortic valve replacement
* Sinus rhythm
* Provide written informed consent

Exclusion Criteria:

* Inclusion in other trial
* Left ventricular ejection fraction less than 0.45
* Presence of any coexisting severe valvular disorder
* Previous cardiac surgery
* Urgent or emergent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Universal definition of perioperative bleeding in adult cardiac surgery | Within 3 days from surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiothoracic Surgery, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Bratt S, Dimberg A, Kastengren M, Lilford RD, Svenarud P, Sartipy U, Franco-Cereceda A, Dalen M. Bleeding in minimally invasive versus conventional aortic valve replacement. J Cardiothorac Surg. 2024 Jun 21;19(1):349. doi: 10.1186/s13019-024-02667-1. PMID 38907320
- [Derived] Kirmani BH, Jones SG, Muir A, Malaisrie SC, Chung DA, Williams RJ, Akowuah E. Limited versus full sternotomy for aortic valve replacement. Cochrane Database Syst Rev. 2023 Dec 6;12(12):CD011793. doi: 10.1002/14651858.CD011793.pub3. PMID 38054555